CLINICAL TRIAL: NCT03984656
Title: Evaluation of the Analgesia by Serratus Plane Block During Pleural Drainage in Intensive Care Unit.
Acronym: SERRATUS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI2018_843_0022
Record Dates: First submitted 2019-06-11; First posted 2019-06-13 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Analgesia; Lidocaine; Intensive Care Unit
Keywords: serratus plane block; analgesia; pleural drainage; lidocaine; intensive care unit
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AL group (Active Comparator): patients will receive a local infiltration of 10 mL Lidocaine without epinephrine 20 mg/mL
  Interventions: Drug: lidocaine treatment
- Serratus group (Experimental): patients will receive ultrasound guided serratus plane block injection of 30 mL Ropivacaine 4.75 mg/mL
  Interventions: Drug: serratus plane block treatment

INTERVENTIONS:
Drug: lidocaine treatment — The index marks the upper edge of the lower rib of the selected intercostal space to avoid the vasculonervous bundle sitting at the lower part of the overlying rib.Non-targeted subcutaneous infiltration is performed in the drainage area with 5 to 10 mL of Lidocaine 20 mg / mL non-adrenaline, plane by plane, with regular aspiration until air or fluid confirming effusion.
  Arms: AL group
Drug: serratus plane block treatment — The Serratus plane block is located at the level of the 5th rib, on the midaxillary line, on the drainage side, ultrasound guided. The block is performed with a 70 mm needle in the ultrasound plane, and the needle is directed postero-inferior, after visualization of the structures from the surface to the depth: dorsal muscle
  * anterior serratus large muscle (serratus anterior)
  * intercostal muscle
  * 4th and 5th ribs
  * pleura A single injection of 30 mL of Ropivacaine 4.75 mg / mL is performed around the Serratus muscle.
  An intravenous injection of 8 mg of Dexamethasone is added to prolong the duration of the block.
  Arms: Serratus group

SUMMARY:
Pleural drainage under local anesthesia is a frequent practice in resuscitation, experienced as an unpleasant and painful event for patients. Pain management is an important issue for early rehabilitation, decrease hospitalisation's cost and shortening the length of stay in intensive care unit (ICU). A new type of locoregional anesthesia called Serratus plane block described by Blanco in 2013 showed a benefit in per and postoperative analgesia in thoracic surgery and carcinologic breast surgery, allowing a decrease in morphine use and an improvement of the patient's general satisfaction. Serratus plane block is a very effective technique in chest wall analgesia, easy and safe to perform, with few complications. No studies to date have evaluated this anesthetic practice in intensive care for pleural drainage. This technique could be used outside the operating room to improve the intensive care patients, who often have heavier pathologies and greater pain, such as patients with chest trauma or patients with cardiac or respiratory disease. The investigators would like to conduct a preliminary study of superiority in the CHU Amiens intensive care unit, to study the interest of the Serratus plane block in comparison with local anesthesia on the management of acute pain during pleural drainage.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years old.
* non-intubated patient with spontaneous ventilation
* free and informed consent of the patient,
* affiliated to a social security scheme
* hospitalized in ICU unit including surgical ICU, cardiothoracic and respiratory ICU or cardiothoracic and respiratory continuous care unit.
* requiring pleural drainage gas or fluid
* conscious patient, not sedated.

Exclusion Criteria:

* patient under the age of 18 years old.
* patient refusal
* under curatorship or deprivation of liberty
* pregnant, parturient or breastfeeding woman
* contraindication to Lidocaine or Ropivacaine
* coagulation disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-06-04 (Actual); Primary Completion 2023-06-04 (Estimated); Study Completion 2023-06-04 (Estimated)

PRIMARY OUTCOMES:
Acute pain intensity measure | at the start of inclusion (H0)
  The assessment of acute pain intensity will be done by numerical pain rating scale during plane-by-plane dissection of pleural drainage (H0). The Numeric Pain Rating Scale (NPRS) is a unidimensional measure of pain intensity in adults. The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain.[3] The common format is a horizontal bar or line. Similar to the VAS, the NPRS is anchored by terms describing pain severity extremes. The most commonly used is the 11-item NPRS. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").

SECONDARY OUTCOMES:
measure of acute pain intensity at rest | at the start of inclusion (H0)
  The assessment of acute pain intensity will be done by numerical pain rating scale during plane-by-plane dissection of pleural drainage (H0). The Numeric Pain Rating Scale (NPRS) is a unidimensional measure of pain intensity in adults. The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain.[3] The common format is a horizontal bar or line. Similar to the VAS, the NPRS is anchored by terms describing pain severity extremes. The most commonly used is the 11-item NPRS. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
measure of acute pain intensity at expiration at the end of pleural drainage | at the start of inclusion (H0)
  The assessment of acute pain intensity will be done by numerical pain rating scale during plane-by-plane dissection of pleural drainage (H0). The Numeric Pain Rating Scale (NPRS) is a unidimensional measure of pain intensity in adults. The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain.[3] The common format is a horizontal bar or line. Similar to the VAS, the NPRS is anchored by terms describing pain severity extremes. The most commonly used is the 11-item NPRS. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Change from baseline (HO) of acute pain at rest following drainage | at one hour after patient inclusion
  The assessment of acute pain intensity will be done by numerical pain rating scale during plane-by-plane dissection of pleural drainage (H0). The Numeric Pain Rating Scale (NPRS) is a unidimensional measure of pain intensity in adults. The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain.[3] The common format is a horizontal bar or line. Similar to the VAS, the NPRS is anchored by terms describing pain severity extremes. The most commonly used is the 11-item NPRS. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Change from baseline (HO) of acute pain at rest following drainage | at 6 hours after patient inclusion
  The assessment of acute pain intensity will be done by numerical pain rating scale during plane-by-plane dissection of pleural drainage (H0). The Numeric Pain Rating Scale (NPRS) is a unidimensional measure of pain intensity in adults. The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain.[3] The common format is a horizontal bar or line. Similar to the VAS, the NPRS is anchored by terms describing pain severity extremes. The most commonly used is the 11-item NPRS. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Change from baseline (HO) of acute pain at rest following drainage | at 24 hours after patient inclusion
  The assessment of acute pain intensity will be done by numerical pain rating scale during plane-by-plane dissection of pleural drainage (H0). The Numeric Pain Rating Scale (NPRS) is a unidimensional measure of pain intensity in adults. The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain.[3] The common format is a horizontal bar or line. Similar to the VAS, the NPRS is anchored by terms describing pain severity extremes. The most commonly used is the 11-item NPRS. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Change from baseline (HO) of acute pain at expiration following drainage | at 1 hour after patient inclusion
  The assessment of acute pain intensity will be done by numerical pain rating scale during plane-by-plane dissection of pleural drainage (H0). The Numeric Pain Rating Scale (NPRS) is a unidimensional measure of pain intensity in adults. The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain.[3] The common format is a horizontal bar or line. Similar to the VAS, the NPRS is anchored by terms describing pain severity extremes. The most commonly used is the 11-item NPRS. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Change from baseline (HO) of acute pain at expiration following drainage | at 6 hours after patient inclusion
  The assessment of acute pain intensity will be done by numerical pain rating scale during plane-by-plane dissection of pleural drainage (H0). The Numeric Pain Rating Scale (NPRS) is a unidimensional measure of pain intensity in adults. The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain.[3] The common format is a horizontal bar or line. Similar to the VAS, the NPRS is anchored by terms describing pain severity extremes. The most commonly used is the 11-item NPRS. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Change from baseline (HO) of acute pain at expiration following drainage | at 24 hours after patient inclusion
  The assessment of acute pain intensity will be done by numerical pain rating scale during plane-by-plane dissection of pleural drainage (H0). The Numeric Pain Rating Scale (NPRS) is a unidimensional measure of pain intensity in adults. The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain.[3] The common format is a horizontal bar or line. Similar to the VAS, the NPRS is anchored by terms describing pain severity extremes. The most commonly used is the 11-item NPRS. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").

CONTACTS AND LOCATIONS:
Overall Officials: Louise Badoux, MD, Principal Investigator — CHU amiens; Stéphanie Malaquin, MD, Principal Investigator — CHU Amiens; Osama Abou Arab, MD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No